CLINICAL TRIAL: NCT05816642
Title: A Prospective Observational Study of Molecular Classification and Circulating Tumor DNA Dynamic Monitoring to Explore Related Factors That Predict the Efficacy of Single Targeted Therapy or Combined With Immunotherapy for Metastatic Renal Cell Carcinoma
Brief Title: Application Circulating Tumor DNA Dynamic Monitoring in Clinical Treatment of Metastatic Renal Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Ruijin Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); West China Hospital (Other); Xiangya Hospital of Central South University (Other); Fudan University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Second Affiliated Hospital of Nantong University (Other); Peking University First Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Zhejiang University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Sir Run Run Shaw Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); The General Hospital of Eastern Theater Command (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The First Affiliated Hospital of University of Science and Technology of China (Other); The Second Hospital of Anhui Medical University (Other); Tongji Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Peking Union Medical College Hospital (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Shanxi Provincial Cancer Hospital (Unknown); Changzhi Medical College (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); The First Affiliated Hospital of Air Force Medicial University (Other); Tang-Du Hospital (Other); Quanzhou First Hospital (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MRCC-China collaboration
Record Dates: First submitted 2022-10-22; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: metastatic renal cell carcinoma; molecular classification; ctDNA dynamic monitoring; targeted therapy; targeted therapy combined with immunotherapy
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib; pazopanib; Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single targeted therapy (Active Comparator): sunitinib or pazopanib
  Interventions: Drug: sunitinib or pazopanib
- targeted therapy combined with immunotherapy (Experimental): Programmed death-ligand 1 Inhibitor combined with axitinib
  Interventions: Drug: PD-1 inhibitor combined with axitinib

INTERVENTIONS:
Drug: sunitinib or pazopanib — Single targeted therapy
  Arms: Single targeted therapy
Drug: PD-1 inhibitor combined with axitinib — targeted therapy combined with immunotherapy
  Arms: targeted therapy combined with immunotherapy

SUMMARY:
Next-Generation Sequencing and whole transcriptome RNA sequencing were used to detect genomic variation and expression in tissues or blood, respectively. The treatment outcome of single targeted therapy or combined with immunotherapy was observed and followed up. Through this study, we intend to achieve RNA molecular classification of Chinese mRCC patients and to evaluate the correlation between ctDNA level, RNA molecular classification and treatment outcome, provide reference for metastatic RCC precise diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with renal cell carcinoma confirmed by pathology, including clear renal cell carcinoma and type I papillary renal cell carcinoma, type II papillary renal cell carcinoma, chromophobe renal cell carcinoma and renal cell carcinoma with sarcomatoid differentiation, etc

  * Have distant metastasis
  * metastatic RCC
  * Eastern Cooperative Oncology Group 0 to 1
  * No obvious abnormality was found in blood routine examination, coagulation and liver and kidney function

Exclusion Criteria:

* • Previously received systematic treatment

  * Failure to obtain baseline tumor tissue / blood samples
  * A history of infection with human immunodeficiency virus, or suffer from other acquired and congenital immunodeficiency diseases, or have a history of organ transplantation, or have a history of organ transplantation
  * A history of allergy to disease treatment drugs
  * During lactation or pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | From drug taken until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 20 months

SECONDARY OUTCOMES:
Objective Response Rate | From drug taken until the date of first documented progression, assessed up to 20 months

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided